CLINICAL TRIAL: NCT03163303
Title: Using Facebook to Address Smoking and Heavy Drinking in Young Adults
Brief Title: Smoking Tobacco and Drinking Study
Acronym: STAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0509092; R34DA041637 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Smoking; Heavy Episodic Drinking
Keywords: Tobacco; Cigarettes; Alcohol; Cessation; Intervention; Young adults; Internet; Social media
MeSH Terms: conditions — Smoking | interventions — Ethanol; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tobacco Status Project (TSP) + Alcohol Intervention (Experimental): Tobacco and alcohol intervention on Facebook and 14-day nicotine patch
  Interventions: Behavioral: Tobacco Status Project + Alcohol Intervention; Drug: nicotine patch
- Tobacco Status Project Intervention (Experimental): Tobacco intervention on Facebook and 14-day nicotine patch
  Interventions: Behavioral: Tobacco Status Project Intervention; Drug: nicotine patch

INTERVENTIONS:
Behavioral: Tobacco Status Project Intervention — 90 days of Facebook messaging, weekly live sessions targeting tobacco use
  Arms: Tobacco Status Project Intervention
Behavioral: Tobacco Status Project + Alcohol Intervention — 90 days of Facebook messaging, weekly live sessions targeting tobacco use and alcohol use
  Arms: Tobacco Status Project (TSP) + Alcohol Intervention
Drug: nicotine patch — 14-day supply of nicotine patch

SUMMARY:
This trial will test the efficacy of a 3-month intervention on Facebook targeting tobacco use and heavy episodic drinking against a 3-month Facebook intervention targeting tobacco use. Both groups will be offered a nicotine patch starter kit. The primary outcome is verified 7-day point prevalence abstinence from smoking at 3, 6, and 12 months.

DETAILED DESCRIPTION:
Participants will be randomized to one of two conditions: (1) a Facebook-delivered intervention addressing tobacco use and heavy episodic drinking, tailored to readiness to quit smoking; or (2) a 3-month Facebook intervention targeting tobacco use. Both interventions will include 12 weeks of Facebook-based messages and activities tailored to participants' readiness to quit smoking.

Assessments will occur at baseline, 3, 6, and 12 months follow-up. Assessments will include measures on smoking and drinking patterns and thoughts about abstinence. All participants who report no past 7-day smoking will be asked to give biochemical verification of smoking status with saliva cotinine test kits that will be mailed to participants.

ELIGIBILITY:
Inclusion Criteria:

* read English
* between 18 and 25 years of age
* indicate they use Facebook "most" (≥ 4) days per week
* have smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* have had at least one heavy drinking episode (5+ for men, 4+ for women) in the past month.

Exclusion Criteria:

* do not read English
* are not between 18 and 25 years of age
* indicate they do not use Facebook "most" (≥ 4) days per week
* have not smoked ≥100 cigarettes in their lives and currently smoke at least 1 cigarette per day on 4 or more days of the week
* have not had at least one heavy drinking episode (5+ for men, 4+ for women) in the past month.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Satre, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Department of Psychiatry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified and transferred to Dr. Chris Yang, expert on social media analytics at Drexel University, for analysis

REFERENCES:
- [Derived] Meacham MC, Ramo DE, Prochaska JJ, Maier LJ, Delucchi KL, Kaur M, Satre DD. A Facebook intervention to address cigarette smoking and heavy episodic drinking: A pilot randomized controlled trial. J Subst Abuse Treat. 2021 Mar;122:108211. doi: 10.1016/j.jsat.2020.108211. Epub 2020 Nov 23. PMID 33509414
- [Derived] Ramo DE, Meacham MC, Kaur M, Corpuz ES, Prochaska JJ, Satre DD. Development of a social media-based intervention targeting tobacco use and heavy episodic drinking in young adults. Addict Sci Clin Pract. 2019 Apr 1;14(1):14. doi: 10.1186/s13722-019-0141-9. PMID 30940206

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the baseline assessment were randomized to the STAND intervention or Tobacco Status Project (TSP) control conditions 1:1 using blocked random assignment sequence generated by the biostatistician. Randomization was stratified by 2 variables known to be related to outcomes: daily smoking status and readiness to quit smoking
Groups:
- Tobacco Status Project + Alcohol Intervention: Tobacco and alcohol intervention on Facebook and 14-day nicotine patch
  Tobacco Status Project + Alcohol Intervention: 90 days of Facebook messaging, weekly live sessions targeting tobacco use and alcohol use
  nicotine patch: 14-day supply of nicotine patch
Period: Overall Study
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Started | 85 | 94
Completed | 85 | 94
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention | Total
Number analyzed (Participants) | 85 | 94 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (2.32) | 22.1 (2.08) | 22.1 (2.20)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 49 | 82
  Male | 40 | 39 | 79
  Transgender or non-binary | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 79 | 92 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 7 | 13
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 66 | 78 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 85 | 94 | 179
Geographic region [Count of Participants; unit: Participants]
  South | 28 | 28 | 56
  West | 21 | 25 | 46
  Midwest | 20 | 24 | 44
  Northeast | 16 | 17 | 33
Number of Cigarettes Smoked in Past 7 days [Mean (Standard Deviation); unit: number of cigarettes] | 76.2 (60.9) | 68.6 (44.7) | 72.6 (53.8)
Usual Number of Cigarettes per Day [Mean (Standard Deviation); unit: cigarettes per day] | 10.1 (6.23) | 10.8 (7.35) | 10.4 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at 3 Months
Description: Point prevalent abstinence was defined as biochemically-verified reports of no smoking in the 7 days prior to the 3 month assessment. Participants reporting no smoking in the past 7 days will be coded as abstinent from cigarettes. Participants with a salivary cotinine level <11 ng/ml, indicating nonsmoking were considered confirmed nonsmokers
Time Frame: 3 months post baseline
Population: Not all participants completed the Month 3 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 69 | 79
Participants | 3 | 4

2. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at 6 Months
Description: Point prevalent abstinence was defined as biochemically-verified reports of no smoking in the 7 days prior to the 6 month assessment. Participants reporting no smoking in the past 7 days will be coded as abstinent from cigarettes. Participants with a salivary cotinine level <11 ng/ml, indicating nonsmoking were considered confirmed nonsmokers
Time Frame: 6 months post baseline
Population: Not all participants completed the Month 6 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 53 | 61
Participants | 0 | 1

3. Primary Outcome: Number of Participants With Reported 7-day Point Prevalence Abstinence at 12 Months
Description: Point prevalent abstinence was defined as biochemically-verified reports of no smoking in the 7 days prior to the 12 month assessment. Participants reporting no smoking in the past 7 days will be coded as abstinent from cigarettes. Participants with a salivary cotinine level <11 ng/ml, indicating nonsmoking were considered confirmed nonsmokers
Time Frame: 12 months post baseline
Population: Not all participants completed the Month 12 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 70 | 81
Participants | 3 | 0

4. Secondary Outcome: Number of Participants With a Reduction in Cigarettes Smoked Over Time
Description: A reduction was defined as the number of cigarettes smoked in past 7 days prior to the assessment by 50% or more compared to baseline number of cigarettes at 3, 6, and 12 month
Time Frame: 3, 6, and 12 months post baseline
Population: Not all participants completed the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
Participants
  Month 3 | 32 | 35
  Month 6 | 35 | 30
  Month 12 | 46 | 46

5. Secondary Outcome: Number of Participants Whom Attempted to Quit Tobacco Use During the Course of Treatment
Description: An attempt was defined by the participants response to the a question as to whether or not they had made an attempt to quit smoking during the course of treatment at the 3, 6, and 12 months post-baseline assessments. Participants who were determined to have made an attempt at least once during the entire course of treatment were scored as yes or no.
Time Frame: 3, 6, and 12 month post-baseline
Population: Not all participants complete the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
Participants | 49 | 45

6. Secondary Outcome: Number of Participant Reporting a Readiness to Quit Tobacco Use Over Time
Description: Readiness to change tobacco use will be assessed with a single-item Readiness Ruler, developed and validated for use with young adult heavy smokers participating in brief intervention and the tobacco item from the Staging Health Risk Assessment (S-HRA) to compare stage of change across tobacco and alcohol use. Plans to limit smoking in next 30 days (or is already). Number of participants ready to change smoking in the next month assessed at 3, 6, and 12 months
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
Participants
  Month 3 | 37 | 27
  Month 6 | 20 | 23
  Month 12 | 34 | 41

7. Secondary Outcome: Average Score on the Thoughts About Abstinence Questionnaire (Smoking)
Description: The Thoughts About Abstinence Questionnaire (TAAS, (Hall et al., 1991) is a 3 item self-report questionnaire that measures: 1) desire to quit smoking, 2) expected success at quitting, 3) expected difficulty of quitting on 10-point Likert scales (e.g., 1=no desire to quit/lowest expectation/lowest level of difficulty to 10 = extreme desire to quit/highest expectation of success/highest expected difficulty) was assessed at baseline.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 85 | 94
score on a scale
  Desire to quit | 6.1 (2.6) | 5.9 (2.5)
  Expected success | 4.6 (2.3) | 5.1 (2.6)
  Expected difficulty | 7.2 (2.4) | 7.1 (2.3)

8. Secondary Outcome: Average Number of Days of Heavy Episodic Drinking (HED) Over Time
Description: HED is defined as the number of days in the past month with 4+ drinks consumed in a a single occasion for women and 5+ drinks for men. HED was assessed at 3, 6 and 12 months.
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
days
  Month 3 | 4.8 (7) | 7.6 (8.2)
  Month 6 | 3.8 (5.5) | 6 (7.8)
  Month 12 | 3.2 (5.2) | 5.6 (7.6)

9. Secondary Outcome: Median Number of Drinks Per Week Over Time
Description: The number of drinks per week was defined as drinks per week in the past 30 days and assessed at the 3,6,and 12 month assessments.
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Median (Inter-Quartile Range); unit: drinks per week
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
drinks per week
  Month 3 | 4 [0 to 12] | 6 [0 to 17]
  Month 6 | 5 [0 to 11] | 7 [0 to 15]
  Month 12 | 1 [0 to 7.8] | 4 [0 to 16]

10. Secondary Outcome: Average Score on the Alcohol Use Disorder Identification Test - Concise (AUDIT-C) Over Time
Description: Misuse of alcohol in the past year was assessed by the AUDIT-C. The AUDIT-C is a brief alcohol screening instrument that reliably identifies persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence) and consists of 3 questions with a total score ranging from 0-12, and generally the higher the score, the more likely it is that a person's drinking is affecting his or her safety. Each AUDIT-C question has 5 answer choices valued from 0 points to 4 points. In men, a score of 4 or more is considered positive, optimal for identifying hazardous drinking or active alcohol use disorders. In women, a score of 3 or more is considered positive. Participants were given this assessment at months 3, 6, and 12.
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
score on a scale
  Month 3 | 3.9 (2.7) | 5 (2.9)
  Month 6 | 3.7 (2.7) | 4.8 (3)
  Month 12 | 3.4 (2.4) | 4.1 (3.1)

11. Secondary Outcome: Alcohol Quit Attempt
Description: Follow-up Drinking Questionnaire will assess the presence and number of 24 hr quit attempts since the last assessment. This assessment will be used to calculate presence of at least one quit attempt in the assessment time period and scored as a yes or no.
Time Frame: 3, 6, and 12 months post-baseline
Population: Data not collected.
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Readiness to Change Alcohol Use Over Time
Description: Readiness to change alcohol use will be assessed with a single-item Readiness Ruler, developed and validated for use with young adult heavy drinkers participating in brief intervention and the alcohol item from the Staging Health Risk Assessment (S-HRA) to compare stage of change across tobacco and alcohol use. Plans to limit drinking in next 30 days (or is already) Proportion of participants ready to change drinking in the next month assessed at 3, 6, and 12 months
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
Participants
  Month 3 | 40 | 42
  Month 6 | 28 | 38
  Month 12 | 42 | 54

13. Secondary Outcome: Average Score on the Thoughts About Abstinence Questionnaire (Heavy Episodic Drinking) Over Time
Description: The Thoughts About Abstinence Questionnaire (TAAS, (Hall et al., 1991) is a 4 item self-report questionnaire that measures: 1) desire to quit heavy episodic drinking, 2) expected success at quitting, 3) expected difficulty of quitting, and 4) confidence in ability to quit on 10-point Likert scales (e.g., 1=no desire to quit; 10 = extremely ...adapted for heavy episodic alcohol use
Time Frame: 3, 6, and 12 months post-baseline
Population: Data not collected.
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Reported Combined Use Using Tobacco or Alcohol Over Time
Description: Timeline Follow-back data will be used to calculate the sum of days using any tobacco or binge drinking in the past month.
Time Frame: 3, 6, and 12 months post-baseline
Population: Not all participants completed the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
Number analyzed (Participants) | 78 | 89
Participants
  Month 3 | 48 | 63
  Month 6 | 36 | 49
  Month 12 | 43 | 52

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Non-serious adverse events were not collected
Arm/Group | Tobacco Status Project + Alcohol Intervention | Tobacco Status Project Intervention
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/94
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Self-reported vaping frequency may have impacted biochemically verified nicotine abstinence validity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03163303/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT03163303/Prot_SAP_001.pdf